CLINICAL TRIAL: NCT06948084
Title: A Randomized Phase II Trial for High-Risk Multiple Myeloma That is Refractory or in First Relapse With Daratumumab, Teclistamab (DT) Versus Daratumumab, Pomalidomide, Dexamethasone (DPd) or Daratumumab, Carfilzomib, Dexamethasone (DKd)
Brief Title: Testing the Investigational Medication Combination of Daratumumab and Teclistamab Compared to the Usual Treatment (Daratumumab, Pomalidomide, Dexamethasone or Daratumumab, Carfilzomib, Dexamethasone) for Patients With High-risk Multiple Myeloma Refractory or in First Relapse
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-02986; NCI-2025-02986 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAA232 (Other: ECOG-ACRIN Cancer Research Group); EAA232 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2025-04-26; First posted 2025-04-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Specimen Handling; Biopsy; carfilzomib; daratumumab; Hyaluronoglucosaminidase; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A Treatment I (DPd) (Active Comparator): Patients receive daratumumab-hyaluronidase SC over 3-5 minutes on days 1, 8, 15, and 22 of cycles 1 and 2, on days 1 and 15 of cycles 3-6, then on day 1 of subsequent cycles. Patients also receive pomalidomide PO on days 1-21 of each cycle, dexamethasone PO or IV on days 1, 8, 15, and 22 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo urine and blood sample collection, bone marrow biopsy, and FDG PET/CT throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Daratumumab and Recombinant Human Hyaluronidase; Drug: Dexamethasone; Procedure: FDG-Positron Emission Tomography; Drug: Pomalidomide
- Arm A Treatment II Option 1 (DKd) (Active Comparator): Patients receive daratumumab-hyaluronidase SC over 3-5 minutes carfilzomib IV on days 1, 2, 8, 9, 15, and 16 of each cycle, and dexamethasone PO or IV on days 1, 2, 8, 9, 15, and 16 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo urine and blood sample collection, bone marrow biopsy, and FDG PET/CT throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Drug: Carfilzomib; Procedure: Computed Tomography; Drug: Daratumumab and Recombinant Human Hyaluronidase; Drug: Dexamethasone; Procedure: FDG-Positron Emission Tomography
- Arm A Treatment II Option 2 (DKd) (Active Comparator): Patients receive daratumumab-hyaluronidase SC over 3-5 minutes on days 1, 8, 15, and 22 of cycles 1 and 2, on days 1 and 15 of cycles 3-6 and on day 1 of subsequent cycles, carfilzomib IV on days 1, 8, and 15 of each cycle, and dexamethasone PO or IV on days 1, 8, 15, and 22 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo urine and blood sample collection, bone marrow biopsy, and FDG PET/CT throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Drug: Carfilzomib; Procedure: Computed Tomography; Drug: Daratumumab and Recombinant Human Hyaluronidase; Drug: Dexamethasone; Procedure: FDG-Positron Emission Tomography
- Arm B (daratumumab, teclistamab) (Experimental): Patients receive daratumumab-hyaluronidase SC over 3-5 minutes on days 1, 8, 15, and 22 of cycles 1 and 2, on days 1 and 15 of cycles 3-6 and on day 1 of subsequent cycles. Patients also receive teclistamab SC on day 2, 4, 8, 15 and 22 of cycle 1, on days 1, 8, 15, and 22 of cycle 2, on days 1 and 15 of cycles 3-6 and then on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo urine and blood sample collection, bone marrow biopsy, and FDG PET/CT throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Daratumumab and Recombinant Human Hyaluronidase; Procedure: FDG-Positron Emission Tomography; Drug: Teclistamab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo urine and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Carfilzomib — Given IV
  Other Names: Carfilnat; CFZ; Kyprolis; PR 171; PR-171; PR171
  Arms: Arm A Treatment II Option 1 (DKd); Arm A Treatment II Option 2 (DKd)
Procedure: Computed Tomography — Undergo FDG PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Daratumumab and Recombinant Human Hyaluronidase — Given SC
  Other Names: DARA Co-formulated with rHuPH20; DARA/rHuPH20; Daratumumab + rHuPH20; Daratumumab and Hyaluronidase; Daratumumab and Hyaluronidase-fihj; Daratumumab and vorhyaluronidase; Daratumumab and Vorhyaluronidase Alfa; Daratumumab with rHuPH20; Daratumumab-rHuPH20; Daratumumab/Hyaluronidase-fihj; Daratumumab/rHuPH20 Co-formulation; Darzalex Faspro; Darzalex/rHuPH20; Darzquro; HuMax-CD38-rHuPH20; Recombinant Human Hyaluronidase Mixed with Daratumumab
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
  Arms: Arm A Treatment I (DPd); Arm A Treatment II Option 1 (DKd); Arm A Treatment II Option 2 (DKd)
Procedure: FDG-Positron Emission Tomography — Undergo FDG PET/CT
  Other Names: FDG; FDG-PET; FDG-PET Imaging
Drug: Pomalidomide — Given PO
  Other Names: 4-Aminothalidomide; Actimid; CC 4047; CC-4047; CC4047; Imnovid; Pomalyst
  Arms: Arm A Treatment I (DPd)
Drug: Teclistamab — Given SC
  Other Names: JNJ 64007957; JNJ-64007957; JNJ64007957; Teclistamab-cqyv; Tecvayli
  Arms: Arm B (daratumumab, teclistamab)

SUMMARY:
This phase II trial compares the effect of the combination of daratumumab-hyaluronidase (daratumumab) and teclistamab to the usual treatment of daratumumab, pomalidomide, dexamethasone or daratumumab, carfilzomib and dexamethasone in treating patients with multiple myeloma that has not responded to previous treatment (refractory) or that has come back after a period of improvement (relapsed). Daratumumab is in a class of medications called monoclonal antibodies. It binds to a protein called CD38, which is found on some types of immune cells and cancer cells, including myeloma cells. Daratumumab may block CD38 and help the immune system kill cancer cells. Teclistamab is a bispecific antibody that can bind to two different antigens at the same time. Teclistamab binds to B-cell maturation antigen, a protein found on some B-cells and myeloma cells, and CD3 on T-cells (a type of white blood cell) and may interfere with the ability of cancer cells to grow and spread. Pomalidomide is in a class of medications called immunomodulatory agents. It works by helping the immune system kill cancer cells and by helping the bone marrow to produce normal blood cells. Dexamethasone is in a class of medications called corticosteroids. It is used to reduce inflammation and lower the body's immune response to help lessen the side effects of chemotherapy drugs. Carfilzomib, a type of proteasome inhibitor, blocks the action of enzymes called proteasomes, which may help keep cancer cells from growing and may kill them. Giving daratumumab and teclistamab may be more effective than the usual treatment of daratumumab, pomalidomide, dexamethasone or daratumumab, carfilzomib and dexamethasone in reducing myeloma cells to undetectable levels in patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether patients with high-risk multiple myeloma (MM) that is refractory or in first relapse randomized to daratumumab and recombinant human hyaluronidase (daratumumab-hyaluronidase) in combination with teclistamab (DT) have superior efficacy measured by minimal residual disease (MRD)-negative status after 6 cycles of therapy compared to investigator's choice of daratumumab-hyaluronidase, pomalidomide and dexamethasone (DPd) or daratumumab-hyaluronidase, carfilzomib and dexamethasone (DKd).

SECONDARY CLINICAL OBJECTIVES:

I. To compare toxicity rates up to 6 cycles and overall on treatment between arms.

II. To compare progression-free and overall survival between arms. III. To evaluate best response per International Myeloma Working Group (IMWG) criteria after 6 cycles and overall on treatment.

IV. To evaluate safety and tolerability.

EXPLORATORY CLINICAL OBJECTIVES:

I. To evaluate treatment exposure and adherence. II. To evaluate time to progression and event free survival. III. To evaluate association of MRD-negative status after 6 cycles with best response per IMWG criteria and time to event outcomes.

EXPLORATORY THROMBOEMBOLISM RISK OBJECTIVES:

I. To estimate cumulative incidence of venous and arterial thromboembolic events.

II. To calculate IMPEDE and SAVED risk scores at baseline and at time of venous thromboembolic event.

III. To validate IMPEDE and SAVED risk stratification models. IV. To describe thromboprophylaxis strategies on treatment and assess the association with venous and arterial thromboembolic events.

V. To estimate incidence of clinically significant (major) bleeding events and assess association with thromboprophylaxis strategy.

VI. To assess the association of venous and arterial thromboembolic events and overall survival.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients are assigned to 1 of 2 treatments per investigator's choice.

Treatment I (DPD): Patients receive daratumumab-hyaluronidase subcutaneously (SC) over 3-5 minutes on days 1, 8, 15, and 22 of cycles 1 and 2, on days 1 and 15 of cycles 3-6, then on day 1 of subsequent cycles. Patients also receive pomalidomide orally (PO) on days 1-21 of each cycle, dexamethasone PO or intravenously (IV) on days 1, 8, 15, and 22 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Treatment II (DKD): Patients are assigned to 1 of 2 options for carfilzomib.

OPTION 1: Patients receive daratumumab-hyaluronidase SC over 3-5 minutes carfilzomib IV on days 1, 2, 8, 9, 15, and 16 of each cycle, and dexamethasone PO or IV on days 1, 2, 8, 9, 15, and 16 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

OPTION 2: Patients receive daratumumab-hyaluronidase SC over 3-5 minutes on days 1, 8, 15, and 22 of cycles 1 and 2, on days 1 and 15 of cycles 3-6 and on day 1 of subsequent cycles, carfilzomib IV on days 1, 8, and 15 of each cycle, and dexamethasone PO or IV on days 1, 8, 15, and 22 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B:

Patients receive daratumumab-hyaluronidase SC over 3-5 minutes on days 1, 8, 15, and 22 of cycles 1 and 2, on days 1 and 15 of cycles 3-6 and on day 1 of subsequent cycles. Patients also receive teclistamab SC on day 2, 4, 8, 15 and 22 of cycle 1, on days 1, 8, 15, and 22 of cycle 2, on days 1 and 15 of cycles 3-6 and then on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Additionally, patients undergo urine and blood sample collection, bone marrow biopsy, and fludeoxyglucose F-18 (FDG) positron emission tomography (PET)/computed tomography (CT) throughout the study.

After completion of study treatment, patients are followed up every 3 months for up to year 2, every 6 months up to year 5 then yearly for up to 10 years from randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥ 18 years of age
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2 (PS 3 allowed if secondary to pain)
* Patient must have an identifiable dominant sequence (clonotype) established based on Adaptive Biotechnologies clonoSEQ® assay
* Patient must have received only one prior line of therapy

  * One prior line of systemic therapy is defined as 1 or more cycles of single agent or combination therapy, as well as a series of treatment regimens administered in a sequential manner (e.g., lenalidomide, bortezomib and dexamethasone induction therapy for 4 cycles followed by autologous stem cell transplantation and then lenalidomide +/- proteasome inhibitor or anti-CD38 monoclonal antibody (mAb) maintenance therapy would be considered 1 line of prior therapy)
  * NOTE: Autologous stem cell transplant is allowed provided the stem cell infusion was > 90 days prior to randomization. Allogeneic stem cell transplantation (SCT) patients are ineligible
* Patient must be diagnosed with relapsed or refractory (RR) multiple myeloma, as defined by disease progression, either an increase in serum or urine M protein of any level, or other evidence of progression biochemical or clinical as specified in the IMWG progression criteria (including disease which becomes non-responsive or progressive on therapy or within 60 days of the last treatment in patients who had achieved a partial response or better on prior therapy)
* Patient must be daratumumab-hyaluronidase (or isatuximab) naïve or daratumumab-hyaluronidase (or isatuximab) sensitive and > 180 days from their last dose of daratumumab-hyaluronidase (or isatuximab) at the time of randomization
* Patient must have high-risk multiple myeloma (HR-MM) as defined by one of the following either at diagnosis or at refractory status or at first relapse:

  * Evidence of deletion 17p by fluorescence in situ hybridization (FISH) testing on bone marrow
  * Evidence of t(4;14) by FISH testing on bone marrow
  * Evidence of t(14;16) by FISH testing on bone marrow
  * Evidence of t(14;20) by FISH testing on bone marrow
  * Evidence of chromosome 1 abnormalities either gain/amp 1q or deletion 1p by FISH testing on bone marrow OR
  * Evidence of non-hyperdiploid karyotype OR
  * Revised International Staging System (R-ISS) stage III beta2 microglobulin ≥ 5.5 mg/L and serum lactate dehydrogenase (LDH) > institutional upper limit of normal (ULN) OR
  * Patient in first relapse and ≤ 24 months from the start of induction for both allogeneic stem cell transplantation (ASCT) eligible or ASCT ineligible patients (regardless of FISH, cytogenetic or RISS stage)
* Patient must have measurable disease as defined by having one or more of the following, obtained within 28 days prior to randomization:

  * Serum M protein ≥ 0.5 g/dL (≥ 5 g/L)
  * Urine M protein ≥ 200 mg/24 hours
  * Serum free light chain (FLC) assay: Involved free light chain level ≥ 10 mg/dL (≥ 100 mg/L) provided serum FLC ratio is abnormal (< 0.26 or > 1.65)
  * Exception: patients without measurable disease in the serum or urine, but with bone or soft tissue plasmacytoma(s) ≥ 2 cm or who have bone marrow plasma cells ≥ 30% are eligible on study
* Patient must have serum protein electrophoresis (SPEP), urine protein electrophoresis (UPEP), and serum FLC assays along with bone marrow biopsy or aspirate performed within 28 days prior to randomization

  * NOTE: UPEP (on a 24 hour collection) is required, no substitute method is acceptable. Urine must be followed monthly if the baseline urine M-spike is ≥ 200 mg/24 hr. If both serum and urine M-components are measurable, both must be followed in order to confirm response
  * NOTE: The serum free light chain test is required to be done at each cycle
* Patient must not have any known allergies, hypersensitivity, or intolerance to corticosteroids, monoclonal antibodies or human proteins, or their excipients (refer to respective package inserts or investigator's brochure), or known sensitivity to mammalian-derived products
* Patients who have received prior systemic therapy for myeloma, including experimental therapy and steroids must have recovered from clinically significant adverse events prior to randomization
* Patient may not be on steroids (prednisone > 40mg/day or equivalent) at the time of randomization
* Patient may have received prior palliative and/or localized radiation, provided that it is completed by the time of randomization
* Absolute neutrophil count (ANC) ≥ 1,000/uL (=< 28 days prior to protocol randomization)
* Untransfused platelet count ≥ 50,000/uL (for patients with ≥ 50% plasma cells in the marrow) and untransfused platelet count > 75,000/uL (for patients with < 50% plasma cells in the marrow) (=< 28 days prior to protocol randomization)
* Untransfused hemoglobin ≥ 8.0 g/dL (=< 28 days prior to protocol randomization)
* Total bilirubin ≤ 1.5 x institutional ULN (upper limit of normal) (=< 28 days prior to protocol randomization)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) ≤ 3.0 × institutional ULN (=< 28 days prior to protocol randomization)
* Calculated creatinine clearance > 30 mL/min (=< 28 days prior to protocol randomization)

  * NOTE: Cockcroft-Gault equation should be used to calculate creatinine clearance
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used

  * All patients of childbearing potential must have a blood test or urine study within 14 prior to randomization to rule out pregnancy. Patients randomized to Arm A and to receive the daratumumab-hyaluronidase, pomalidomide, dexamethasone (DPd) regimen must also have a second pregnancy test within 24 hours prior to the first dose of pomalidomide and agree to ongoing pregnancy testing while on protocol treatment
  * A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patient must not expect to conceive or father children by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study and for 5 months after the last dose of protocol treatment for patients on Arm B and for 3 months after the last dose of protocol treatment for patients on Arm A. In addition, patients randomized to Arm A and receive the daratumumab-hyaluronidase, pomalidomide, dexamethasone (DPd) regimen must also agree to register to the mandatory Risk Evaluation and Mitigation Strategies (REMS®) program and be willing and able to comply with the requirements of the REMS program. All patients must not breastfeed while on protocol treatment and for patients on Arm B they must not breastfeed for an additional 5 months after the last dose of protocol treatment
* Patient may have primary plasma cell leukemia (pPCL), secondary plasma cell leukemia (sPCL) or extramedullary myeloma (EMM)
* Patient must not have evidence of active or untreated central nervous system (CNS) positive MM. Patients with prior CNS involvement are eligible provided they had demonstrated evidence of CNS disease resolution by imaging and/or 2 consecutively negative cerebrospinal fluid (CSF) samples for the presence of plasma cells
* Patient must not have active autoimmune disease
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of randomization are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patients with a history of chronic obstructive pulmonary disease (COPD) must have forced expiratory volume in 1 second (FEV1) testing done within 28 days prior to randomization and the forced expiratory volume in 1 second (FEV1) must be >= 50% of predicted normal
* Patient must not have moderate or severe persistent asthma within 2 years prior to randomization

  * NOTE: Patients who currently have controlled intermittent asthma or controlled mild persistent asthma are eligible
* Investigator must declare the intended chemotherapy regimen at the time of randomization should their patient be randomized to Arm A from the two options

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-29 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease (MRD) negativity | After 6 cycles of treatment (cycle length = 28 days), assessed at 6 months
  Will be determined by the Adaptive Biotechnologies clonoSEQ assay result. Analysis will be performed using Cochran-Mantel-Haenszel (CMH) test, stratified on prior anti-CD38 antibody therapy and investigator's choice of therapy if assigned to Arm A. MRD-negative status requires both MRD negativity and achievement of complete response. Will be summarized using descriptive statistics by treatment arm with two-sided exact binomial 80% confidence intervals (CI), Clopper-Pearson. The corresponding CMH odds ratio (OR) estimate with an 80% CI, and p-value will be reported. Logistic regression will be used to assess the treatment effect within subgroups including but not limited to age 70 status, prior anti-CD38 antibody therapy and high-risk by fluorescence in situ hybridization status.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 6 cycles (cycle length = 28 days) and overall assessed up to 10 years
  Will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) and classified by Medical Dictionary for Regulatory Activities (MedDRA) system organ class. Maximum grade toxicity by AE type will be tabulated. Summaries (count and percentages) will be reported by AE type by arm.
Incidence of grade 3 or higher hematologic and/or non-hematologic AEs | Up to 6 cycles (cycle length = 28 days) and overall assessed up to 10 years
  Will be graded according to the NCI CTCAE and classified by MedDRA system organ class. Maximum grade toxicity by AE type will be tabulated. Summaries (count and percentages) will be reported by AE type by arm. Rates of maximum grade 3 or higher (including grade 5) non-hematologic, hematologic and overall toxicity will be calculated along with 90% CIs. AEs will be further analyzed by arm in subsets of serious AEs per protocol, lethal AEs and treatment-emergent AEs status.
Progression-free survival (PFS) | From randomization until the earlier of progression or death due to any cause, assessed up to 10 years
  PFS will be estimated in the treated population using the Kaplan-Meier method and compared between arms using the stratified log-rank test. Stratified cox proportional hazards (PH) regression will be used to produce the treatment hazard ratio (HR) along with the 90% CI, provided PH assumption is valid. Sensitivity analyses excluding untreated patients will be conducted.
Overall survival (OS) | From randomization to death due to any cause, assessed up to 10 years
  OS will be estimated in the treated population using the Kaplan-Meier method and compared between arms using the stratified log-rank test. Stratified cox PH regression will be used to produce the treatment HR along with the 90% CI, provided PH assumption is valid. Sensitivity analyses excluding untreated patients will be conducted.
Response rates | After 6 cycles of treatment (cycle length = 28 days) and overall, assessed up to 10 years
  Will be reported by treatment arm. Rates of stringent complete response (CR) or better, very good partial response (VGPR) or better and partial response (PR) or better will be computed along with 90% CIs in all treated patients. Stratified CMH test will be used to test the difference in VGPR or better rates between arms. Sensitivity analyses excluding untreated patients will be conducted.

OTHER OUTCOMES:
Event-free survival | From randomization until the earlier of non-protocol therapy, progression, or death due to any cause, assessed up to 10 years
Time to progression | From randomization to time of documented progression or censored at date of last disease evaluation if alive or death not due to disease progression, assessed up to 10 years
Duration of treatment | From randomization to treatment end, or censored at the date of last treatment, assessed up to 10 years
Cumulative dose intensity | Up to 24 months (cycle length = 28 days)
  Will be defined as the sum of all doses taken across all cycles. Will be characterized using descriptive statistics.
Number of dose modifications (DM) | Up to 6 cycles (cycle length = 28 days) and overall, assessed up to 10 years
  The number of DMs, DM status (planned versus unplanned) and reason for DM by cycle and overall treatment will be characterized using descriptive statistics. Reasons off treatment and every DM will also be tabulated.
Relative dose intensity | Up to 6 cycles (cycle length = 28 days) and overall, assessed up to 10 years
  Will be defined as the dose received as percentage of planned dose of each cycle. Will be characterized using descriptive statistics.
Incidence of venous thromboembolism (VTE) | Up to 10 years
  The cumulative incidence of VTE overall and within dichotomized risk groups will be assessed using Fine and Gray model with and without adjustment for age and competing risk of death. To assess the impact of thrombosis on survival, incidence of VTE will be treated as a time-dependent covariate in Cox PH regression models of survival follow-up. Computed HR and 90% CI will be reported. Additionally, landmark (LM) analyses with patients alive classified by occurrence of VTE after 6 cycles of treatment based on Kaplan Meier from that timepoint will be conducted.
Incidence of arterial thrombotic events (ATE) | Up to 10 years
  The cumulative incidence of ATE overall and within dichotomized risk groups will be assessed using Fine and Gray model with and without adjustment for age and competing risk of death. To assess the impact of thrombosis on survival, incidence of ATE will be treated as a time-dependent covariate in Cox PH regression models of survival follow-up. Computed HR and 90% CI will be reported. Additionally, LM analyses with patients alive classified by occurrence of ATE after 6 cycles of treatment based on Kaplan Meier from that timepoint will be conducted.
Incidence of clinically significant bleeding events | Up to 10 years
  Will be assessed according to concurrent thromboprophylaxis type and dose.
Venous thromboembolism risk | At baseline and at time of VTE, assessed up to to 24 months
  IMPEDE and SAVED risk scores will be calculated. Patients will be classified into 3 risk groups (low, intermediate, high) and dichotomized (low vs. intermediate-high) based on IMPEDE risk score while patients will be classified into 2 risk groups (low and high) based on SAVED risk score. Descriptive statistics will be used to characterize IMPEDE and SAVED risk variables and scores. The accuracy of IMPEDE and SAVED risk models will be assessed based on positive predictive value.
Thromboprophylaxis | Up to 24 months (cycle length = 28 days)
  Descriptive statistics (count and percentages) will be used to characterize thromboprophylaxis strategies (type and dose).
Impact of MRD-negative status on PFS and OS | After 6 cycles (cycle length = 28 days)
  Kaplan Meier plots will be produced by MRD-negative status as defined in this study. Alternative definitions of MRD-negative status and MRD levels will also be assessed. MRD assessment will also be evaluated in the context of disease response based on standard International Myeloma Working Group (IMWG) criteria. The proportion of patients with marrow MRD-negative status will be cross-tabulated with IMWG response categories (PR, VGPR, CR, stringent complete response [sCR]). Sensitivity analyses excluding untreated patients will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Muhamed Baljevic, Principal Investigator — ECOG-ACRIN Cancer Research Group

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm